CLINICAL TRIAL: NCT05852509
Title: Digital Health Physical Activity Program for Older Family Care Partners of Patents With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-4757; K23AG073471 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Caregiver Burden
Keywords: heart failure; older adults; family caregivers; digital health; physical activity
MeSH Terms: conditions — Heart Failure; Caregiver Burden; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPA4You group (Experimental): Participants in the TPA4You group will be given an overview of the TPA4You program and PA exercise safety instructions. HF-FCPs will receive 28 PA sessions delivered by the coach over 12 weeks. The coached sessions will taper from 3 days/week (weeks 1-4) to 2 days/week (weeks 5-12) but exercise on 3 days/week will be recommended throughout. Participants will receive tailored motivational text messages every other day to encourage daily exercise and wearing the Fitbit.
  Interventions: Behavioral: TPA4You
- Attention control group (Other): Participants will be given booklets, provided by the NIA, AHA, and National Alliance for Caregiving that include content about self-care for FCPs' health and well-being, but not specific to PA or exercise. Participants will receive text messages every other day to encourage them to wear the Fitbit device, and to provide friendly greetings and reminders of upcoming survey data collection.
  Interventions: Behavioral: Attention control group

INTERVENTIONS:
Behavioral: TPA4You — TPA4You integrates technology components in the form of video-conferencing (e.g., Zoom) with a health coach, wearable sensor (e.g., Fitbit), and personalized text messaging into a package to (a) tailor physical activity (PA) prescriptions based on the family care partners of persons with heart failure (HF-FCP)'s feedback and individual wearable sensor data, (b) provide tailored PA coaching sessions using video-conferencing, and (c) motivate daily exercise using text messages.
  Arms: TPA4You group
Behavioral: Attention control group — Participants will be given booklets, provided by the NIA, AHA, and National Alliance for Caregiving, that include content about self-care for FCPs' health and well-being, but not specific to PA or exercise. Participants will receive text messages every other day to encourage them to wear the Fitbit device, and to provide friendly greetings and reminders of upcoming survey data collection.
  Arms: Attention control group

SUMMARY:
The purpose of the Aim 3 study is to conduct a pilot randomized controlled trial to assess feasibility and preliminary effects of the TPA4You intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years
* Involved in caring for a household member aged 50 years or older with the New York Heart Association Class II, III or IV HF
* Provide at least 8 hours/week of unpaid care for the past 3 months
* Physically able to engage in structured exercise such as walking, and upper body resistance exercises
* Engage in < 30 min of moderate-intensity exercise on fewer than 3 days per week
* Able to read, speak, and comprehend 5th grade English
* Own a smartphone
* Reachable by telephone, text messaging, and email
* Have a 6x6ft space fit for physical activity in the place of residence

Exclusion Criteria:

* Medical or functional conditions precluding participation in the physical activity (PA) components of the intervention (e.g., inability to walk one block or climb stairs without chest pain, shortness of breath, dizziness; history of falls; or serious or unstable cardiovascular or pulmonary disease)
* Cognitive impairment (Telephone Interview for Cognitive Status [TICS] score < 25)
* Inability to use technology
* Participation in a PA intervention in the previous 6 months
* Current participation in a PA or behavior change trial
* Physical activity unpreparedness ('Yes' to any questions 1-4 the Physical Activity Readiness Questionnaire [PAR-Q]. If participants respond 'yes' to any questions 5-7, we will ask follow-up questions.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Daily physical activity counts | 6 months
  Daily physical activity counts will be measured using the Fitbit Inspire 2 wearable wristband which is an accelerometer-based activity tracker. Total PA counts will be downloaded from the Fitbit app.

SECONDARY OUTCOMES:
Sedentary activity | 6 months
  Sedentary activity will be measured using the Fitbit Inspire 2 wearable wristband which is an accelerometer-based activity tracker. The data will be downloaded from the Fitbit app. Sedentary activity is defined as less than 100 counts/min.
Physical function | 6 months
  30-Second Chair Stand Test will be used to assess lower-body strength. The coach will explain the test to participants and measure performance. Participants will sit squarely in a stable chair with arms crossed over chest, and, with a straight back rise to a full standing position without use of hands, return to the seated position and repeat for 30 seconds.
Depression | 6 months
  Depression will be measured using the Center for Epidemiological Studies Depression Scale (CES-D), a 20-item questionnaire rated on a 4-point Likert scale ranging from 0 to 3 (higher scores = worse depressive symptom).
Anxiety | 6 months
  Anxiety will be measured using the State Trait Anxiety Index, a 20-item questionnaire rated on a 4-point scale with total scores from 1 to 80 (higher scores = worse anxiety symptom).
Stress | 6 months
  Stress will be measured using the Perceived Stress Scale (PSS), a 10-item questionnaire rated on a 5-point Likert scale ranging from 0 to 4 (higher scores = worse stress).
Caregiving self-efficacy | 6 months
  Caregiving self-efficacy will be measured using the Revised Scale for Caregiving Self-Efficacy (RSCSE), a 15-item questionnaire rated on an 11-point scale ranging from 0 to 100 (higher scores = better self-efficacy).
Health related quality of life | 6 months
  Health related quality of life (HRQoL) will be measured using the Short Form 36 version 2,a 36-item questionnaire with 2 domains (physical and psychological health) (higher scores = better HRQoL).
Usability of TPA4You | 6 months
  Self-reported ease of use and usability of TPA4You will be measured with the refined 20-item Health Information Technology (IT) Usability Evaluation Scale (Health-ITUES) (higher scores = better usability).
Total sleep time | 4 months
  Total sleep time will be measured using the Fitbit Inspire 2 wearable wristband and collected from the Fitbit app.
Wake after sleep onset | 6 months
  Wake after sleep onset will be measured using the Fitbit Inspire 2 wearable wristband and collected from the Fitbit app.
Sleep efficiency | 6 months
  Sleep efficiency will be measured using the Fitbit Inspire 2 wearable wristband and collected from the Fitbit app.

CONTACTS AND LOCATIONS:
Overall Officials: Dawon Baik, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baik D, Coats H, Reeder B, Allen LA, Jankowski C. Digital health physical activity coaching for older family caregivers of persons with heart failure - TPA4You: Protocol for a pilot randomized controlled trial. Contemp Clin Trials Commun. 2026 Jan 20;49:101604. doi: 10.1016/j.conctc.2026.101604. eCollection 2026 Feb. PMID 41631240